CLINICAL TRIAL: NCT03241368
Title: Multicenter, Prospective, Study Comparing PillCam® Crohn's Capsule Endoscopy (CE) to Ileocolonoscopy (IC) Plus MRE for Detection of Active Crohn's Disease (CD) in the Small Bowel and Colon in Subjects With Known CD and Mucosal Disease
Brief Title: Clinical Study Comparing PillCam® Crohn's Capsule Endoscopy to Ileocolonoscopy (IC) Plus MRE for Detection of Active CD in the Small Bowel and Colon in Subjects With Known CD and Mucosal Disease.
Acronym: BLINK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COVSBCC0549
Record Dates: First submitted 2017-07-24; First posted 2017-08-07 (Actual); Results first posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2019-10

CONDITIONS: Crohn Disease
Keywords: Irritable Bowel Disease; IBD; Mucosal Disease; Crohn's; Inflammatory Bowel Disease
MeSH Terms: conditions — Crohn Disease; Irritable Bowel Syndrome; Inflammatory Bowel Diseases | interventions — Capsule Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MRE, Patency Capsule (if needed), CE, and IC (Other): Single-arm study, which includes MRE procedure, Patency Capsule Procedure (if needed), PillCam Crohn's Capsule Endoscopy Procedure and Ileocolonoscopy procedure.
  Interventions: Device: Capsule Endoscopy

INTERVENTIONS:
Device: Capsule Endoscopy — At baseline subject will under the PillCam Crohn's Capsule Procedure
  Other Names: PillCam Crohn's® Capsule

SUMMARY:
This study will evaluate the efficacy of capsule endoscopy (CE) versus ileocolonoscopy (IC) plus MRE for detection of active Crohn's disease (CD) in the small bowel in subjects with known CD and mucosal disease.

The primary objective of the study is to assess the accuracy of CE versus IC plus MRE for detecting active CD, by visualizing the small bowel and colon in subjects with known CD and mucosal disease.

There will be assessment of mucosal disease activity at baseline. Patient satisfaction questionnaire will be completed at baseline.

DETAILED DESCRIPTION:
This is a multicenter, prospective, study, evaluating the efficacy of CE versus IC plus MRE for detecting active Crohn's Disease (CD) in the small bowel and colon in subjects with known CD and mucosal disease.

A screening visit will be performed within 30 days prior to baseline procedures to assess pre-procedure eligibility. At this visit the following assessments will be performed: Informed Consent, Inclusion/Exclusion Criteria, Demographics, Montreal Classification, Medical History, Previous GI procedures, Surgical history, Laboratory tests and pregnancy tests.

At baseline, subjects with known CD on routine evaluation (e.g. history, physical exams, labs) and a recent history of mucosal disease (within the last 2 years and diagnosis based on radiologic, endoscopic, or histologic findings) OR subjects with known CD and active disease based on clinical judgment based on symptoms, laboratory data or other clinical information will undergo Magnetic Resonance Enterography (MRE), Capsule Endoscopy (CE) and Ileocolonoscopy (IC), to assess presence or absence of CD across the small and large bowel. Also, at baseline the following assessments will take place: Laboratory tests, Pregnancy test, Concomitant medications, Patient satisfaction questionnaire and Adverse Events (AE).

Subjects will be exited from the study once all Baseline Procedures have been completed and AEs resolved.

All CE videos, IC videos and MRE images will be evaluated by central readers.

The planned number of subjects is 352. Subjects will be enrolled at up to 40 sites in the United States, Israel, and Austria. Study duration is expected to be up to approximately 1.5 years. The expected duration of each subject's participation is approximately 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent.
* Subject is ≥ 18 years of age
* Subject is willing and able to comply with all aspects of treatment and evaluation schedule.
* Subject has known CD and a recent history (within last 2 years) of mucosal disease (based on radiologic, endoscopic, or histologic evidence) OR known CD and active disease, based on clinical judgment based on symptoms, laboratory data or other clinical information.

Exclusion Criteria:

* Subject has indeterminate, ulcerative, antibiotic-associated colitis.
* Subject has stool positive for ova and parasite and for Clostridium difficile toxins within 3 months prior to enrollment.
* Subject with other known infectious cause of abdominal symptoms.
* Subject with clinical evidence of renal disease with the past 6 months, defined as estimated glomerular filtration rate (GFR) outside the normal reference range.
* Subject with known history of intestinal obstruction or current obstructive symptoms, such as severe abdominal pain with accompanying nausea or vomiting, based on investigator judgment.
* Subject with a diagnosis of gastroparesis or small bowel or large bowel dysmotility.
* Subject with suspected or known bowel obstruction, stricture (defined as unequivocal proximal upstream dilation equal ≥ 2.5 cm), or fistula.
* Subject has used non-steroidal anti-inflammatory drugs including aspirin, two times per week, during the 4 weeks preceding enrollment. Low dose aspirin regimens (≤ 100 mg daily) are acceptable and not exclusionary.
* Subject suffers from any condition, such as swallowing problems, that precludes compliance with study and/or device instructions.
* Subject with cardiac pacemaker or other implanted electromedical device.
* Subject has an allergy or other known contraindication to the medications used in the study.
* Subject is pregnant (documented by a positive pregnancy test) or is actively breast-feeding.
* Subject is considered to be a part of a vulnerable population (eg. prisoners or those without sufficient mental capacity).
* Subject has a known contraindication to MRE or IC.
* Subject has participated in a drug or device research study within 30 days of enrollment that may interfere with the subject's safety or ability to participate in the study.
* Subject has any medical condition that would make it unsafe for them to participate, per Investigator's discretion
* Subject with ileostomy or colostomy, history of total or subtotal colectomy (including those with ileosigmoidostomy, and ileorectostomy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Bruining, MD, Principal Investigator — Mayo
Locations (26):
- United States (24):
  - University of South Alabama, Mobile, Alabama
  - Mayo Clinic (Scottsdale, AZ), Scottsdale, Arizona
  - Encore Borland Groover Clinical Research, Jacksonville, Florida
  - Children's Center for Digestive Healthcare, Atlanta, Georgia
  - Loyola University - Chicago, Maywood, Illinois
  - Indiana University, Indianapolis, Indiana
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - University of Kansas, Kansas City, Kansas
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic (Rochester, MN), Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Atlantic Health (Morristown), Morristown, New Jersey
  - Asheville Gastroenterology Associates, PA, Asheville, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Digestive Disease Specialists Inc., Oklahoma City, Oklahoma
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Carilion Clinic, Roanoke, Virginia
  - Virginia Gastroenterology Institute, Suffolk, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Allgemeines Krankenhaus - Universitatskliniken Wein, Vienna, Austria
- Sheba Medical Center, Tel Litwinsky, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bruining DH, Oliva S, Fleisher MR, Fischer M, Fletcher JG; BLINK study group. Panenteric capsule endoscopy versus ileocolonoscopy plus magnetic resonance enterography in Crohn's disease: a multicentre, prospective study. BMJ Open Gastroenterol. 2020 Jun;7(1):e000365. doi: 10.1136/bmjgast-2019-000365. PMID 32499275

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 187 subjects signed consent. Per the protocol, a subject was not considered "enrolled" until consent was signed and subject met inclusion/exclusion criteria. Of the 187 who signed consent, 158 were considered "enrolled" per the protocol. 29 were "screen failures", i.e. they signed informed consent, but ended up failing inclusion/exclusion.
Pre-assignment Details: Of the 187 subjects who signed informed consent, 29 failed inclusion/exclusion criteria and were exited from the study. Criteria included labs, which caused some subjects to wash out at this early phase. This left us with 158 subjects. For various reasons, 39 additional subjects were exited prior to all imaging procedures being completed.
Groups:
- MRE, Patency Capsule (if Needed), CE, and IC: Subjects will undergo MRE, patency capsule (if necessary), CE, and IC procedures.
  If MRE shows evidence of a stricture, subject must undergo a Patency procedure prior to CE. If patency not confirmed by MRE or patency capsule, subject is discontinued from study.
  Subjects will perform bowel preparation and follow a detailed dietary regimen for CE and IC procedures. Between 45 and 75 minutes after final polyethylene glycol (PEG) ingestion, subject will swallow the PillCam Crohn's Capsule. Adequate boosts will be administered, as necessary. Subjects will be allowed to leave clinic after 'Alert 2' is received and if capsule is not yet excreted. Subjects leaving prior to excretion will be instructed to disconnect the recorder at excretion or battery failure (whichever is first).
  After CE procedure (either same or following day), subject will undergo IC. If IC is done the following day, subject will stay on clear liquid diet (or NPO (nothing by mouth), per physician discretion).
Period: Overall Study
Arm/Group | MRE, Patency Capsule (if Needed), CE, and IC
Started | 158
Completed | 119
Not Completed | 39
Not completed — MRE Stricture or Patency Capsule Failure | 25
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 6
Not completed — Withdrawal by Subject | 6
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Per-protocol analysis set, included subjects who underwent MRE, CE, and IC (and could be evaluated for CD activity) with no major protocol deviations (violations that may have significant impact on outcomes) and did not meet the following: subject withdraw; capsule remained in stomach or small bowel for entire procedure; system technical failure
Groups:
- MRE, Patency Capsule (if Needed), CE, and IC: Subjects will undergo MRE, patency capsule (if necessary), CE, and IC procedures.
  If MRE shows evidence of a stricture, subject must undergo a Patency procedure prior to CE. If patency cannot be confirmed through MRE or patency capsule will be discontinued from the study.
  Subjects will perform bowel preparation and follow a detailed dietary regimen for CE and IC procedures. Between 45 and 75 minutes after final PEG ingestion, subject will swallow the PillCam Crohn's Capsule. Adequate boosts will be administered, as necessary. Subjects will be allowed to leave clinic after 'Alert 2' is received and if capsule is not yet excreted. Subjects leaving prior to excretion will be instructed to disconnect the recorder at excretion or battery failure (whichever is first).
  After CE procedure (either same or following day), subject will undergo IC. If the IC is done the following day, subject will stay on clear liquid diet (or NPO, per physician's discretion for sedation).
Arm/Group | MRE, Patency Capsule (if Needed), CE, and IC
Number analyzed (Participants) | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 96
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 2
  United States | 95
  Israel | 2
BMI [Mean (Standard Deviation); unit: kg/m²] | 28.82 (7.36)

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of CE Versus IC Plus MRE for Detecting Active Crohn's Disease (CD), by Visualizing the Small Bowel and Colon in Subjects With Know CD and Mucosal Disease.
Description: Central readers will be used to read all videos/images and analyses will be based on these results. A consensus panel will be used if there are discrepancies in results between modalities at baseline. Capsule endoscopy and IC results will be read by gastroenterologists and MRE results will be read by radiologists.
  Scores used will be Lewis Score, Simple Endoscopic Score for Crohn's Disease Index (SES-CD) Score and Magnetic Resonance Index of Activity (MaRIA) Score
Time Frame: Baseline
Population: Per-protocol analysis set, includes subjects who underwent MRE, CE, and IC (and could be evaluated for CD activity) who had no major deviations (violations that may have significant impact on outcomes) and did not meet following criteria:
  * Subject withdraws
  * Capsule remained in stomach or small bowel for entire procedure
  * Technical failure
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | MRE, Patency Capsule (if Needed), CE, and IC
Number analyzed (Participants) | 99
percentage of participants
  Sensitivity CE Overall | 94 [86 to 98]
  Sensitivity MRE + IC Overall | 100 [95 to 100]
  Specificity CE Overall | 74 [55 to 87]
  Specificity MRE + IC Overall | 22 [10 to 41]
Statistical Analysis 1: Comparison: MRE, Patency Capsule (if Needed), CE, and IC; This was a 1-arm, non-powered study. Sensitivity, Specificity, Positive Predictive Value (PPV) and Negative Predictive Value (NPV) was estimated for each treatment group, along with the 95% confidence interval. The difference between treatment groups in Sensitivity and Specificity was compared; Test type: Other — Comparative - This purpose of this study is to evaluate performance of the PillCam Crohn's capsule [referred to as capsule endoscopy (CE)] as compared to IC with MRE; p = 0.125, McNemar; Exact McNemar's test

2. Secondary Outcome: Specificity, Negative Predictive Value, and Positive Predictive Value for Active CD in the Small Bowel and Colon by CE as Compared to IC Plus MRE.
Description: as for outcome 1
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | MRE, Patency Capsule (if Needed), CE, and IC
Number analyzed (Participants) | 99
percentage of participants
  Specificity | 74 [55 to 87]
  Negative Predictive Value (NPV) | 83 [64 to 94]
  Positive Predictive Value (PPV) | 91 [82 to 96]

3. Secondary Outcome: Sensitivity, Specificity, Negative Predictive Value and Positive Predictive Value for Active CD in Designated Bowel Segments (Proximal Small Bowel Terminal Ileum, and Colon) by Capsule Endoscopy as Compared to IC Plus MRE
Description: as for outcome 1
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | MRE, Patency Capsule (if Needed), CE, and IC
Number analyzed (Participants) | 99
percentage of participants
  Sensitivity CE Proximal Small Bowel (PSB) | 97 [82 to 100]
  Sensitivity MRE PSB | 71 [53 to 84]
  Specificity CE PSB | 87 [76 to 93]
  Specificity MRE PSB | 66 [54 to 76]
  NPV CE PSB | 98 [90 to 100]
  NPV MRE PSB | 83 [71 to 91]
  PPV CE PSB | 77 [62 to 88]
  PPV MRE PSB | 49 [35 to 63]
  Sensitivity CE Terminal ilium (TI) | 94 [84 to 99]
  Sensitivity MRE + IC TI | 98 [89 to 100]
  Specificity CE TI | 82 [66 to 91]
  Specificity MRE + IC TI | 37 [23 to 53]
  NPV CE TI | 91 [76 to 98]
  NPV MRE + IC TI | 93 [68 to 100]
  PPV CE TI | 88 [76 to 94]
  PPV MRE + IC TI | 68 [57 to 78]
  Sensitivity CE Colon | 83 [62 to 94]
  Sensitivity IC Colon | 91 [72 to 99]
  Specificity CE Colon | 88 [77 to 94]
  Specificity IC Colon | 89 [79 to 95]
  NPV CE Colon | 93 [84 to 98]
  NPV IC Colon | 97 [88 to 100]
  PPV CE Colon | 70 [51 to 84]
  PPV IC Colon | 75 [56 to 88]

4. Secondary Outcome: Patient Satisfaction
Description: Patient preference of which procedure they preferred (CE, IC or MRE plus IC)
Time Frame: After completion of final procedure, either the same day or by the next business day following procedure completion.
Population: Subjects who completed the satisfaction questionnaire and underwent all 3 procedures MRE, CE, and IC and could be evaluated for overall active CD at baseline (i.e., a modified intent-to-treat (mITT).
  population).
Measure: Count of Participants; unit: Participants
Arm/Group | MRE, Patency Capsule (if Needed), CE, and IC
Number analyzed (Participants) | 118
Participants
  Preferred PillCam CE | 64
  Preferred IC | 43
  Preferred MRE + IC | 11

ADVERSE EVENTS:
Time Frame: 6 weeks plus 30 days - Events will be collected for all enrolled subjects with the start of baseline imaging procedures (MRE) and end 14 days following completion of the IC procedure. Subjects with Adverse Event (AE) 14 days following the IC procedure will be followed for 30 days or until event resolves, whichever comes first.
Arm/Group | MRE, Patency Capsule (if Needed), CE, and IC
All-Cause Mortality (participants affected / at risk) | 0/119
Serious Adverse Events (participants affected / at risk) | 7/119
Other Adverse Events (participants affected / at risk) | 11/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MRE, Patency Capsule (if Needed), CE, and IC (N=119)
Abdominal pain (Gastrointestinal disorders) | 1
Crohn's Disease (Gastrointestinal disorders) | 3
Complication of device removal (General disorders) | 1
Clostridium difficile infection (Infections and infestations) | 1
Serum sickness (Immune system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MRE, Patency Capsule (if Needed), CE, and IC (N=119)
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Infusion site extravasation (General disorders) | 1
Oesophageal candidiasis (Infections and infestations) | 1
Staphylococcal skin infection (Infections and infestations) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Haemoglobin decreased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Emotional distress (Psychiatric disorders) | 1
Fatigue (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-16): https://cdn.clinicaltrials.gov/large-docs/68/NCT03241368/Prot_SAP_000.pdf